CLINICAL TRIAL: NCT02238379
Title: Oxytocin Pilot: Oxytocin and Face Perception
Brief Title: Intranasal Oxytocin Administration and the Neural Correlates of Social and Non-Social Visual Perception
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Anna Freud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1309012677
Record Dates: First submitted 2014-09-04; First posted 2014-09-12 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Social Perception
Keywords: Intranasal oxytocin; Social perception; EEG/ERP
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Oxytocin (Experimental): Each participant will receive both the oxytocin nasal spray in one visit AND the placebo nasal spray in another visit (randomized) in this design.
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Each participant will receive both the oxytocin nasal spray in one visit AND the placebo nasal spray in another visit (randomized) in this design.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oxytocin — 24 International Units of Oxytocin in a Nasal Spray
  Other Names: Pitocin
  Arms: Oxytocin
Other: Placebo — Placebo will contain all ingredients except the active oxytocin in the Nasal Spray.
  Arms: Placebo

SUMMARY:
The objective of this study is to investigate the effects of oxytocin on social behavior and brain activity using EEG and the event-related potential (ERP) technique. The value of EEG is its high temporal specificity, enabling precision in the timing of social behavior to be addressed. In order to elicit social responses in the human brain, a variety of social and emotional visual stimuli will be presented during EEG recording, namely infant and adult faces and houses. Brain responses after intranasal oxytocin will then be compared with placebo, to examine the effect of intranasal oxytocin on central nervous system activity. We hypothesize that intranasal oxytocin will enhance the neural response to social stimuli (infant and adult faces) but not to non-social stimuli (houses).

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-64
* Good medical health
* Ability to understand and speak English

Exclusion Criteria:

* Pregnancy
* Medical Illnesses: Moderate or severe acute or chronic medical illnesses (e.g. cardiac disease, diabetes, epilepsy, influenza).
* Cardiovascular risk factors: History of hypertension with baseline blood pressure above 140 mm Hg (systolic) over 90 mm Hg (diastolic). Also any history of syncope and/or baseline blood pressure below 100 mm Hg (systolic).
* CNS disease: Known history of brain abnormalities (e.g., neoplasms, subarachnoid cysts), cerebrovascular disease, infectious disease (e.g., abscess), other central nervous system disease, or history of head trauma which resulted in a persistent neurologic deficit or loss of consciousness > 3 minutes.
* Medication status: Individuals on stable doses of a neuroleptic and/or an antidepressant medication for at least the past 6 weeks will be allowed to participate in this study. The use of other psychotropic medications will not be allowed. Females taking contraceptive hormones will not be able to participate in the study.
* A history of seizures or current use of anticonvulsants; history of head injury with loss of consciousness

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda C Mayes, MD, Principal Investigator — Yale University; Helena JV Rutherford, PhD, Study Director — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxytocin First, Then Placebo: Each participant will receive both the oxytocin nasal spray in one visit AND the placebo nasal spray in another visit (randomized) in this design.
  Oxytocin: 24 International Units of Oxytocin in a Nasal Spray
- Placebo First, Then Oxytocin: Each participant will receive both the oxytocin nasal spray in one visit AND the placebo nasal spray in another visit (randomized) in this design.
  Placebo: Placebo will contain all ingredients except the active oxytocin in the Nasal Spray.
Period: Overall Study
Arm/Group | Oxytocin First, Then Placebo | Placebo First, Then Oxytocin
Started | 12 | 14
Completed | 11 | 14
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: 1 participant was lost to follow up for their placebo visit (determined after blind was broken).
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (3) | 23 (3) | 24 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Amplitude Social
Description: The investigators will analyze the amplitude (i.e., size) of visually elicited event-related potential (ERP) components to the social stimuli (infant and adult faces). This assessment will be completed after administration of the intervention (oxytocin) and the placebo to compare the neural response. The investigators hypothesize that the intervention will modulate the amplitude of the neural response to social stimuli given its previously identified role in social interactions, most likely increasing the size of the ERPs.
Time Frame: Duration of 30 minutes
Population: 1 participant was lost to follow-up (did not complete placebo); 1 participant's data was lost (removed then from placebo and oxytocin arms); for LPP analysis, 1 participant was a statistical outlier and removed from oxytocin and placebo arms
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 24 | 24
microvolts
  N170 Infant Distress Faces | -3.72 (2.81) | -3.55 (2.64)
  N170 Infant Neutral | -3.28 (2.55) | -3.30 (2.94)
  N170 Adult Distress | -3.70 (2.72) | -3.27 (2.64)
  N170 Adult Neutral | -3.23 (2.48) | -2.87 (2.33)
  P300 Infant Distress Face | 0.94 (1.26) | 0.50 (1.21)
  P300 Infant Neutral Face | 1.10 (1.47) | 0.55 (1.34)
  P300 Adult Distress Face | 0.65 (1.22) | 0.39 (0.91)
  P300 Adult Neutral Face | 0.52 (1.38) | 0.61 (1.09)
  LPP Infant Distress Face: number analyzed (Participants) | 23 | 23
  LPP Infant Distress Face | -0.56 (1.53) | -0.50 (0.94)
  LPP Infant Neutral Face: number analyzed (Participants) | 23 | 23
  LPP Infant Neutral Face | -0.24 (1.40) | -0.54 (1.51)
  LPP Adult Distress Face: number analyzed (Participants) | 23 | 23
  LPP Adult Distress Face | -0.38 (1.33) | -0.57 (1.40)
  LPP Adult Neutral Face: number analyzed (Participants) | 23 | 23
  LPP Adult Neutral Face | -0.71 (1.49) | -0.40 (1.27)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; N170 Analysis; Test type: Superiority or Other; p = .003, ANOVA — Main Effect of Emotion; Spray (Oxytocin, Placebo) by Face Type (Infant, Adult) by Emotion (Distress, Neutral) by Hemisphere (Left, Right) ANOVA
Statistical Analysis 2: Comparison: Oxytocin vs Placebo; N170 Analysis; Test type: Superiority or Other; p = .034, ANOVA — Main Effect of Face Type; Spray (Oxytocin, Placebo) by Face Type (Infant, Adult) by Emotion (Distress, Neutral) by Hemisphere (Left, Right) ANOVA
Statistical Analysis 3: Comparison: Oxytocin vs Placebo; P300 Analysis; Test type: Superiority or Other; p = .03, ANOVA — Main Effect of Face Type; Spray Type (Oxytocin, Placebo) by Face Type (Infant, Adult) by Emotion (Distress, Neutral) ANOVA
Statistical Analysis 4: Comparison: Oxytocin vs Placebo; P300 Analysis; Test type: Superiority or Other; p = .03, ANOVA — Spray Type by Face Type Interaction; Spray Type (Oxytocin, Placebo) by Face Type (Infant, Adult) by Emotion (Distress, Neutral) ANOVA
Statistical Analysis 5: Comparison: Oxytocin vs Placebo; LPP Analysis; Test type: Superiority or Other; p > .22, ANOVA — No Main Effects or Interactions; Spray Type (Oxytocin, Placebo) by Face Type (Infant, Adult) by Emotion (Distress, Neutral) ANOVA

2. Primary Outcome: Amplitude Non-Social
Description: The investigators analyze the amplitude (i.e., size) of visually elicited event-related potential (ERP) components to the non-social stimuli (houses). This assessment will be completed after administration of the intervention (oxytocin) and the placebo to compare the neural response. The investigators hypothesize that there will be no difference between the intervention and placebo during the non-social condition on the amplitude of the ERPs.
Time Frame: Duration of 30 minutes
Population: 1 participant was lost to follow-up (did not complete placebo); 1 participant's data was lost (removed then from placebo and oxytocin arms)
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 24 | 24
microvolts
  N170 House | -1.15 (1.71) | -1.15 (1.35)
  P300 House | 1.21 (1.47) | 0.86 (0.91)
  LPP House | -0.58 (1.12) | -0.32 (1.06)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; N170 Analysis; Test type: Superiority or Other; p > .14, ANOVA — No Main Effects or Interactions; Spray Type (Oxytocin, Placebo) and Hemisphere (left, right) ANOVA
Statistical Analysis 2: Comparison: Oxytocin vs Placebo; P300 Analysis; Test type: Superiority or Other; p > .17, t-test, 2 sided — No difference between Spray Types; Paired samples t-test comparing Spray Type (Oxytocin vs Placebo)
Statistical Analysis 3: Comparison: Oxytocin vs Placebo; LPP Analysis; Test type: Superiority or Other; p > .27, t-test, 2 sided — No difference between Spray Types; Paired samples t-test comparing Spray Type (Oxytocin vs Placebo)

3. Primary Outcome: Latency Social
Description: The investigators analyze the latency (i.e., efficiency of processing) of visually elicited ERP components to the social stimuli (infant and adult faces). This assessment will be completed after administration of the intervention (oxytocin) and the placebo to compare the neural response. The investigators hypothesize that there will be more efficient processing (i.e., earlier latency) of ERPs during the social condition following administration of the intervention relative to the placebo condition.
Time Frame: Duration of 30 minutes
Population: 1 participant was lost to follow-up (did not complete placebo); 1 participant's data was lost (removed then from placebo and oxytocin arms); for LPP analysis, 1 participants were statistical outliers and removed from oxytocin and placebo arms for N170 latency analysis
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 23 | 23
milliseconds
  N170 Infant Distress | 164 (8) | 164 (10)
  N170 Infant Neutral | 163 (9) | 161 (9)
  N170 Adult Distress | 164 (10) | 163 (12)
  N170 Adult Neutral | 161 (9) | 161 (11)
  Left N170 Infant Distress | 165 (9) | 166 (10)
  Right N170 Infant Distress | 164 (8) | 162 (9)
  Left N170 Infant Neutral | 165 (11) | 163 (10)
  Right N170 Infant Neutral | 161 (7) | 160 (9)
  Left N170 Adult Distress | 166 (11) | 165 (14)
  Right N170 Adult Distress | 162 (9) | 161 (9)
  Left N170 Adult Neutral | 163 (10) | 162 (13)
  Right N170 Adult Neutral | 159 (8) | 160 (10)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Only relevant for N170; Test type: Superiority or Other; p = .006, ANOVA — Main Effect of Emotion; Spray Type (Oxytocin, Placebo), Face Type (Infant, Adult), Emotion (Neutral, Distressed), and Hemisphere (left, right) ANOVA
Statistical Analysis 2: Comparison: Oxytocin vs Placebo; Only relevant for N170; Test type: Superiority or Other; p = .01, ANOVA — Main Effect of Hemisphere; [statistical method as in outcome 3, analysis 1]

4. Primary Outcome: Latency Non-Social
Description: The investigators will analyze the latency (i.e., efficiency of processing) of visually elicited ERP components to the non-social stimuli (houses). This assessment will be completed after administration of the intervention (oxytocin) and the placebo to compare the neural response. The investigators hypothesize that there will be no difference between the intervention and placebo on ERP latency measures in the non-social condition.
Time Frame: Duration of 30 minutes
Population: 1 participant was lost to follow-up (did not complete placebo); 1 participant's data was lost (removed then from placebo and oxytocin arms); 2 participants were statistical outliers and removed from oxytocin and placebo arms for N170 latency analysis
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 23 | 23
milliseconds
  Left N170 House | 171 (13) | 174 (14)
  Right N170 House | 166 (9) | 169 (13)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Only relevant for N170; Test type: Superiority or Other; p = .03, ANOVA — Main Effect of Spray; Spray (oxytocin, placebo) by Hemisphere (left, right) ANOVA
Statistical Analysis 2: Comparison: Oxytocin vs Placebo; Only relevant for N170; Test type: Superiority or Other; p = .008, ANOVA — Main Effect of Hemisphere; Spray (oxytocin, placebo) by Hemisphere (left, right) ANOVA

5. Secondary Outcome: Depression
Description: The investigators will assess depression by employing the Beck Depression Inventory (Beck et al., 1961). Specifically addressing whether the level of depression symptomatology in participants and whether this is associated with the neural correlates of social and non-social perception during both intervention and placebo visits. It is not yet known the extent to which variation in depression symptoms are associated with this methodology, although prior research has suggested depression modulates the neural response to social cues. This measure includes a question regarding suicidal ideation and therefore it is acknowledged there may be a safety issue in response to the questionnaire. Scores range from 0-63, with higher scores indicating greater levels of depression (scores 29+ indicates severe depression).
Time Frame: Within 20 minutes of study visit commencing
Population: Only participants included that have ERP data to analyze (excluding participant lost to follow-up and data loss)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale | 4.00 (6.06) | 4.33 (5.75)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Superiority or Other; p = .05, correlation

6. Secondary Outcome: Smoking
Description: Participants will complete a CO breathalyzer and the Fagerstrom Test for Nicotine Dependence (Heatherton, Kozlowski, Frecker, & Fagerstrom, 1991) to assess smoking behavior. These measures are included to characterize the sample in respect of substance use.
Time Frame: Within 30 minutes of study visit commencing
Population: 1 participant was lost to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 26 | 25
Participants
  FTND indicated smoking status | 1 | 0
  CO indicated smoking status | 0 | 0

7. Secondary Outcome: Anxiety
Description: The investigators will assess anxiety using the State-Trait Anxiety Inventory (Spielberger et al., 1970). Specifically, it will be explored whether participant anxiety symptoms are associated with the neural correlates of social and non-social perception during both intervention and placebo visits. It is not yet known the extent to which variation in anxiety symptoms are associated with this methodology, although prior research has suggested anxiety modulates the neural response to social cues. Scores range from 20-80 and a higher score on both state and trait measures indicate higher levels of anxiety. A potential clinical cut off has been proposed for participants scoring over 39-40 as being high anxious.
Time Frame: Within 20 minutes of study visit commencing
Population: Only participants included that have ERP data to analyze (excluding participant lost to follow-up and data loss)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale
  State Anxiety | 31.54 (10.67) | 35.50 (11.27)
  Trait Anxiety | 30.58 (10.11) | 30.79 (7.82)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Superiority or Other; p = .05, correlation

8. Secondary Outcome: Stress
Description: The investigators will measure current levels of stress by using the Perceived Stress Scale (Cohen et al., 1983). It is not yet known the extent to which variation in perceived stress is associated with this methodology, but it is anticipated stress will be associated with levels of depression and anxiety in the sample. The PSS consists of 14 items, with scores ranging from 0 to 42, with higher scores indicating higher levels of perceived stress. A score of 21+ is considered to indicate that participants have higher than average stress.
Time Frame: Within 20 minutes of study visit commencing
Population: Only participants included that have ERP data to analyze (excluding participant lost to follow-up and data loss)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale | 17.54 (8.28) | 18.13 (8.23)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Superiority or Other; p = .05, correlation

9. Secondary Outcome: Early Experience
Description: The investigators will employ the Parental Bonding Instrument (Parker, Tupling, & Brown, 1979) to assess the early relationship experiences participants have with their caregivers. Existing research employing intranasal oxytocin suggests that the quality of early relationships may impact the strength of any modulation of brain or behavior by oxytocin administration and therefore this variable will be included in the analyses in support of this hypothesis. There are 12 items that capture parental care and 13 items that capture parental overprotection. Items are scored on a 4-point likert scale from "very like" to "very unlike". The PBI is typically scored by identifying optimal (High Care Scores, Low Protection Scores) and less optimal (Low Care Scores, Low Protection Scores) scores on the mother and father subscales (NB: protection refers to overprotection). For the care items, scores can range from 0 to 36; for overprotection items, scores can range from 0 to 39.
Time Frame: Within 20 minutes of study visit commencing
Population: Only participants included that have ERP data to analyze (excluding participant lost to follow-up and data loss); 1 participant did not know their father and did not complete the measure for paternal assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale
  Maternal Care Score | 30.13 (6.69) | 29.50 (6.79)
  Paternal Care Score: number analyzed (Participants) | 23 | 23
  Paternal Care Score | 27.74 (8.67) | 28.13 (8.95)
  Maternal Protectiveness Score | 13.71 (8.01) | 13.75 (8.51)
  Paternal Protectiveness Score: number analyzed (Participants) | 23 | 23
  Paternal Protectiveness Score | 11.91 (8.30) | 10.91 (9.34)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Superiority or Other; p = .05, correlation

10. Secondary Outcome: Number of Participants Endorsing Substance Use
Description: The investigators will employ the ASI Lite (McLellan, Luborsky, Woody, & O'Brien, 1980) to assess for current substance use. This measure is included to characterize the sample in respect of substance use; however the ASI Lite did not provide a measure of substance dependance and therefore we report the data from the Mini International Neuropsychiatric Interview substance dependance module (Sheehan et al., 1998) to provide a specific indication of the presence of absence of substance dependance.
Time Frame: Within 30 minutes of study visit commencing
Population: 1 participant lost to follow-up; count of participants where substance dependence indicated
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 11 | 14
Participants | 0 | 2

11. Secondary Outcome: Number of Participants Testing Positive for Alcohol Use Following a Breathalyzer
Description: Participants will complete an alcohol breathalyzer to characterize the alcohol use status of the sample.
Time Frame: Within 30 minutes of study visit commencing
Population: 1 participant lost to follow-up; data indicates number of participants with alcohol in their system
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 11 | 14
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Oxytocin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25

LIMITATIONS AND CAVEATS:
Small sample size limiting the interpretations of ERP differences between oxytocin and placebo conditions and individual difference measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes